CLINICAL TRIAL: NCT03867630
Title: The Effect of Additional Transforaminal Epidural Blocks in Percutaneous Epidural Neuroplasty With Wire Type Catheter in Lumbar Foraminal Stenosis Patients
Brief Title: The Effect of Additional Transforaminal Epidural Blocks in Percutaneous Epidural Neuroplasty
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Jong Bum Choi, Assistant Professor, Ajou University School of Medicine
Other Study IDs: AJIRB-MED-OBS-18-554
Record Dates: First submitted 2019-03-05; First posted 2019-03-08 (Actual); Last update posted 2019-05-13 (Actual); Status verified 2019-05

CONDITIONS: Lumbar Spinal Stenosis
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Runoff Group: Runoff group are the patients whose images were shown root shadow by contrast media.
- Nonrunoff-Transforaminal group: Nonrunoff-Transforaminal group are the patients whose images are not shown root shadows by contrast media, so additional transforaminal blocks are done.
  Interventions: Procedure: Transforaminal Block
- Nonrunoff-NonTransforaminla group: Nonrunoff-NonTransforaminal group are the patients whose images are not shown root shadows by contrast media, but no additional transforaminal blocks are done.

INTERVENTIONS:
Procedure: Transforaminal Block — Epidural block via neural foramen of lumbar spine
  Groups: Nonrunoff-Transforaminal group

SUMMARY:
Percutaneous epidural neuroplasty (PEN) is an effective interventional treatment for radicular pain. But in some cases with wire catheter like Racz catheter, contrast runoffs were not shown to the foramen. This study will show that contrast runoff will affect the results of PEN and in cases which contrast runoff are not shown, additional transforaminal epidural blocks will affect the results of PEN by reviewing medical record, retrospectively.

DETAILED DESCRIPTION:
Medical records will be investigated in cases of PEN with wire type catheter from May 2016 to August 2018. About one hundred cases will be enrolled. Analysis will be performed. It will be compared 1) Success rate of Runoff group and Nonrunoff group in lumbar spine, 2) Success rate of Runoff group and Nonrunoff-NonTransforaminal group in lumbar spine. 3) Success rate of Runoff group with nonrunoff-transforaminal group and Nonrunoff-NonTransforaminal group in lumbar spine. 4) Success rate of Nonrunoff-Transforaminal group and Nonrunoff-NonTransforaminal group in lumbar spine.

ELIGIBILITY:
Inclusion Criteria:

* 20 to 80 years old
* Patients with a herniated disc, spinal stenosis
* Patients with chronic low back pain and lower extremity pain who did not respond to lumbar epidural steroid injections
* Patients who are performed percutaneous epidural neuroplasty with wire type catheter.

Exclusion Criteria:

* Incomplete medical record
* Contraindication to percutaneous epidural neuroplasty

Ages: 20 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Medical records will be reviewed retrospectively about 100 patients with chronic low back pain and lower extremity pain who did not respond to lumbar epidural steroid injections. As the next stage of treatment, percutaneous epidural neuroplasty with a wire type catheter is performed. The patient's symptoms, neurological examination, and imaging studies were evaluated to make a diagnosis. Patients 20 to 80 years old with a herniated disc, spinal stenosis are included. Percutaneous epidural neuroplasty using a wire type catheter was done, and patients had regular follow-up visits until 1 months after the neuroplasty.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-05-10 (Estimated); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Success rate of three groups | 1 month
  Success rate of three groups(Runoff group, Nonrunoff-foraminal group, Nonrunoff-Nonforaminal group) will be compared each other. Success is defined as a 50% or greater reduction in pain score on the pre-procedural Visual Analogue Scale(VAS) score.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gil HY, Lee SY, Min SK, Kim JE, Lee HS, Jeong HW, Park B, Choung J, Choi JB. The effect of additional transforaminal epidural blocks on percutaneous epidural neuroplasty with a wire-type catheter: A retrospective observational study. Medicine (Baltimore). 2019 Dec;98(50):e18233. doi: 10.1097/MD.0000000000018233. PMID 31852086